CLINICAL TRIAL: NCT07195578
Title: Three Dimensional Puzzle (3D Puzzle) Game Applied to Geriatric Individuals Cognitive Skills and Impact on Life Engagement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, MERVE AKPINAR YILMAZ, ÖĞRETİM GÖREVLİSİ, Eskisehir Osmangazi University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 224S415
Record Dates: First submitted 2025-09-10; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Geriatric Care
Keywords: Keywords: Elderly, cognitive skills, life engagement, puzzle game, geriatric nursing

STUDY DESIGN:
Intervention Model Description: The study was completed with a total of 40 individuals, 20 in the intervention group and 20 in the control group, at the Bolvadin Nursing Home affiliated with the Afyonkarahisar Provincial Directorate of Family and Social Services. The 3D puzzle game was administered to the individuals in the intervention group, three days a week, for a total of 10 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): 3D PUZZLE APPLICATION FOR 10 WEEKS
  Interventions: Other: Three Dimensional Puzzle Game (3D puzzle)
- Control group (No Intervention): CONTINUING ROUTINE INTERNAL ACTIVITIES

INTERVENTIONS:
Other: Three Dimensional Puzzle Game (3D puzzle) — Individuals in the intervention group were exposed to the 3D puzzle game three days a week for a total of 10 weeks. Three-dimensional puzzle figures, ranging in size from 20 to 50 pieces, were used in 30 sessions, each with a different figure.
  Arms: Intervention group

SUMMARY:
Title: Three Dimensional Puzzle (3D Puzzle) Game Applied to Geriatric Individuals Cognitive Skills and Impact on Life Engagement* Objective: The research is a randomized controlled experimental study with a pre-test-post-test design conducted to evaluate the effects of a three-dimensional puzzle (3D puzzle) game applied to geriatric individuals on cognitive skills and life engagement.

Materials and Methods: The study was completed with a total of 40 individuals, 20 in the intervention group and 20 in the control group, at the Bolvadin Nursing Home affiliated with the Afyonkarahisar Provincial Directorate of Family and Social Services. The 3D puzzle game was administered to the individuals in the intervention group, three days a week, for a total of 10 weeks. Three-dimensional puzzle figures, with pieces ranging from 20 to 50, were administered in 30 sessions, each with a different figure. The Standardized Mini Mental Test was used in the sample selection process. Research data were collected using the "Introductory Information Form," the "Montreal Cognitive Assessment Scale," the "Life Engagement Scale," the "Individual Tracking Form," and the "Three-Dimensional Puzzle Assessment Form." Data were analyzed using the Shapiro-Wilk, Kolmogorov-Smirnov, Chi-square (χ²) independent samples t-test, dependent samples t-test, Mann-Whitney U, and Wilcoxon rank-order tests.

Results: At the end of the three-dimensional puzzle game, a significant increase in the mean MOCA score of the geriatric individuals in the intervention group was observed (p<0.001). In terms of the cognitive dimensions of the MOCA scale, significant improvements were observed in the "Attention and Concentration" cognitive dimension (p=0.006) and the "Visual Construction Skills" cognitive dimension (p=0.001) in the intervention group. Following the 3D puzzle game, it was determined that the mean Life Engagement Scale score of the geriatric individuals in the intervention group showed a significant increase (p=0.012).

Conclusion: The study determined that the 3D puzzle game applied to geriatric individuals had a positive effect on cognitive skills and life engagement.

ELIGIBILITY:
Inclusion Criteria:

Age 65 and over

* Agree to participate in the study
* Can speak and understand Turkish
* Can read and write
* Can understand and comply with simple commands
* Individuals without upper extremity motor dysfunction (hand tremors, paralysis, etc.)
* Individuals who scored 24 or higher on the Standardized Mini Mental State Examination

Exclusion Criteria:

- • Individuals with a psychiatric diagnosis that could affect mental status, such as major depression

* Individuals with a chronic neurological disorder [dementia, cerebrovascular accidents (excluding transischemic attacks), epilepsy, Parkinson's disease, mental retardation]
* Individuals with severe hearing and vision problems
* Individuals with complex illnesses such as malignancy
* Individuals with upper extremity motor dysfunction (hand tremors, paralysis, etc.)
* Individuals whose routine treatment plan has been changed
* Individuals participating in another ongoing study

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-01-24 (Actual); Study Completion 2025-07-24 (Actual)

PRIMARY OUTCOMES:
Mean MOBID score of geriatric individuals | Outcome assessed after 10 weeks of intervention
  In terms of the cognitive dimensions of the MOCA scale, significant improvements were observed in the "Attention and Concentration" cognitive dimension (p=0.006) and the "Visual Construction Skills" cognitive dimension (p=0.001) in the intervention group.

CONTACTS AND LOCATIONS:
Locations (1):
- Bolvadin Nursing Home Directorate, Afyonkarahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Fissler, P., Küster, O. C., Loy, L. S., Laptinskaya, D., Rosenfelder, M. J., von Arnim, C. A., & Kolassa, I. T. (2017). Jigsaw Puzzles as Cognitive Enrichment (PACE)-the effect of solving jigsaw puzzles on global visuospatial cognition in adults 50 years — https://doi.org/10.36720/csji.v5i1.426
- See also: Related Info — https://doi.org/10.37036/ahnj.v9i2.454